CLINICAL TRIAL: NCT00308373
Title: Effects of Elevated Free Fatty Acids on Endogenous Glucose Production in People With and Without Type 2 Diabetes Mellitus
Brief Title: Effects of Fats on Blood Glucose in People With and Without Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1104-04; DK29953-FFA/TZD
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

INTERVENTIONS:
Drug: Metformin vs Thiazolidinedione (Pioglitazone)

SUMMARY:
People with type 2 diabetes mellitus (earlier known as maturity onset diabetes mellitus) have high blood levels of sugar and fat. This study is being done to determine if excessive sugar entering the blood in people with type 2 diabetes mellitus is caused by excessive fat. We will also evaluate how the anti-diabetic medications, pioglitazone and metformin taken by mouth work to control blood sugar in people with diabetes.

DETAILED DESCRIPTION:
The ultimate goal of this application is to determine the cause(s) of type 2 diabetes mellitus. The role of the liver in the evolution of type 2 diabetes has not been as extensively studied as that of muscle. This has been, in part, due to the inherent difficulty of measuring hepatic insulin action in humans under physiologic conditions. Plasma free fatty acids (FFA) can cause insulin resistance in non-diabetic humans and are commonly elevated in people with type 2 diabetes. We will re-examine the mechanism(s) by which elevated FFA cause hepatic insulin resistance in non-diabetic humans, will determine whether elevated FFA alter insulin induced suppression of endogenous glucose production (EGP) in diabetic humans and if so, whether this is due to changes in glycogenolysis and/or gluconeogenesis. We will also seek to determine whether treatment with a pioglitazone (a thiazolidinedione) blunts or prevents FFA induced hepatic (and extrahepatic) insulin resistance in people with type 2 diabetes and whether the effects of FFA on insulin action are influenced by gender. We will examine if use of thiazolidinediones reduces cortisol production by changing the overall activity of 11 beta hydroxysteroid dehydrogenase type 1. We will also investigate whether use of thiazolidinediones alters objectively measured breathing or sleepiness in people with type 2 diabetes.

ELIGIBILITY:
Forty-two (21 women, 21 men) diabetic and 31 (16 women, 15 men) matched non-diabetic volunteers will be recruited. Diabetic volunteers whose HbA1c is 7-9% if managed with diet alone or 6.5-8.5% if on either a sulfonylurea or metformin will be eligible for the study. Diabetic and non-diabetic subjects will be healthy and matched for age, gender, and body mass index. Individuals with a body mass index less than 19 or greater than 44 kg/m2 will be excluded from study to avoid potential confounding effects that may result from extreme leanness or obesity. Subjects greater than age 35 years of age will be eligible for study. Subjects less than 35 years will not be studied in order to minimize the possibility of type 1 diabetes. Healthy diabetic subjects will mean that the participant has no history of a) proliferate retinopathy; b) significant nephropathy, (i.e., plasma creatinine > 1.4 mg/dl in women and 1.5 mg/dl in men, and/or proteinuria); c) symptomatic autonomic neuropathy; d) clinically significant atherosclerotic vascular disease (e.g., history of MI or angina); e) a known systemic illness. To ensure subjects are healthy, following informed written consent, subjects will undergo a history and physical examination; blood will be collected for a complete blood count and chemistry group; urine will be collected to insure there is no evidence of infection or clinically significant proteinuria. Body composition (including percent fat, visceral fat, hepatic fat, and lean body mass) will be measured in eligible subjects in the GCRC body composition core using DEXA and a multiple cut CT scan. (Diabetic volunteers will again undergo body composition studies in Part 2 of the protocol, after about 4 months of therapy. Please see below)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2004-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Rizza, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States